CLINICAL TRIAL: NCT05230394
Title: Randomized Control Trial to Compare Patient Outcomes Following Unattended Polysomnography Versus In-lab Polysomnography for Sleep Apnea and Comorbid Sleep Disorders
Brief Title: Patient Outcomes in Unattended and In- Lab Polysomnography
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Issues
Sponsor: Cerebra Medical (Industry)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SDC Study
Record Dates: First submitted 2021-12-30; First posted 2022-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea; Hypersomnia
MeSH Terms: conditions — Sleep Apnea Syndromes; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Level 1 In Lab Polysomnography (Experimental)
  Interventions: Diagnostic Test: Attended Polysomnography in the Lab
- Level 2 In Home Polysomnography (Experimental)
  Interventions: Diagnostic Test: Unattended Polysomnography in the Home

INTERVENTIONS:
Diagnostic Test: Attended Polysomnography in the Lab — Using standard Level 1 polysomnography
  Arms: Level 1 In Lab Polysomnography
Diagnostic Test: Unattended Polysomnography in the Home — Using Cerebra's Prodigy system
  Arms: Level 2 In Home Polysomnography

SUMMARY:
This randomized controlled study will directly evaluate whether unattended polysomnography (level 2 sleep study) in individuals referred for sleep apnea or hypersomnia, including those with comorbidities of insomnia and sleep-related movement disorders, provides similar patient outcomes when compared to level 1 sleep studies.

DETAILED DESCRIPTION:
Individuals referred to the Sleep Disorder Centre with a major complaint of snoring or, apneas or hypersomnia, with at least one additional minor concern of snoring, apneas, restless leg syndrome or insomnia, will be considered for entry into the study. Using a randomized controlled trial design, study participants will be randomly assigned to either the intervention group who will undergo a full unattended polysomnography (level 2 home sleep study) using the Prodigy portable wireless sleep monitor or in-lab polysomnography (level 1 sleep study). Other aspects of care including the clinical assessment will be equivalent between groups. A randomly assigned sleep specialist physician will make treatment recommendations to the patient based on the sleep study results and determine the need for a subsequent testing (including repeat sleep studies) as part of each patient encounter. Physicians participating in the study will receive an introduction to the Odds Ratio Product (ORP) and training on its diagnostic potential. Diagnostic confidence using a 5 point Likert scale from 10% (very unsure) to 90% (very confident) will be assessed after each sleep study review.

ELIGIBILITY:
Inclusion Criteria:

* referral for major concern of "snoring" or "apnea" or "hypersomnia" with additional minor concerns of "snoring", "apneas" "restless leg syndrome" or "insomnia"
* willing to undergo a sleep study

Exclusion Criteria:

* referrals where parasomnias, respiratory failure, narcolepsy listed as concerns
* comorbid congestive heart failure, ischemic heart disease, arrhythmia, stroke, chronic obstructive pulmonary disease/respiratory failure, patients with a BMI 50 kg/m2
* undergone a previous sleep study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Outcomes of Sleep Questionnaire | 4 months
  Total Score scale ranges from 5-20, with higher scores representing better functioning
Change in Epworth Sleepiness Scale | 4 months
  Scale ranges from 0-24, with higher scores representing more sleepiness
Continuous Positive Airway Pressure (CPAP) Adherence | 4 months
  Percent of nights with CPAP > 4 hours/night
Change in Calgary Sleep Apnea Quality of Life Index | 4 months
  Total score ranges from 1-7, with a greater score indicating a lower effect of OSA on quality of life
Rating of Physician Diagnostic Confidence | within 4 weeks of sleep study, after patient assessment by physician
  Likert scale rating performed by physicians to assess confidence in diagnosis from data provided by the two systems, scale from 1-5 with higher values reflecting greater confidence
Rating of Patient Satisfaction | Measured in morning following their sleep study
  Likert scale rating of patient satisfaction for their sleep study experience, ranges from 1-7 with higher values reflecting greater satisfaction
Cost between Level 1 and Level 2 tests based on equipment, facility, supply costs, and technician and physician service fees | After study conclusion, an average of up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No